CLINICAL TRIAL: NCT00360919
Title: Assessing the Presence of Casomorphins in Human Plasma After Dairy Ingestion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: WCCR-01
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Food Habits
Keywords: casomorphin; cheese; craving; casein; milk
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Cheese
  Interventions: Behavioral: cheese ingestion
- B (Placebo Comparator): Fruits and vegetables
  Interventions: Behavioral: cheese ingestion

INTERVENTIONS:
Behavioral: cheese ingestion — On study day 1, approximately half of the participants will consume a breakfast of fruits and vegetables, whereas the other half of participants will consume a meal consisting of 9 oz. of cheese.
  Blood samples will be collected from participants immediately prior to consumption of the meals, and then again at regular intervals for up to 8 hours following the meals.
  At least 3 days later, participants will return for study Day 2. The participants will receive the second meal. Blood samples will then be collected immediately prior to consumption of the test meal and for up to 8 hours after the meal.

SUMMARY:
This purpose of this study is to perform a pilot investigation to determine if opioid peptides such as casomorphin can be detected in human plasma after cheese ingestion.

DETAILED DESCRIPTION:
Cheese is one of the most commonly craved foods, suggesting the possibility of opiate activity, as has been demonstrated with other craved foods, particularly chocolate. Like other dairy products, cheese contains casein, which is the major protein in cow's milk. This is unlike human milk, in which the primary protein is whey. Casein includes αs1-, αs2-, β- , and κ-casein, with αs1 and β forms predominating. Human and bovine casein molecules are cleaved during digestion to release opioid peptides that are believed to have biological properties relevant to infant physiology and behavior. Specifically, β-casein is cleaved to form β-casomorphins. Like other opiate agonists, β-casomorphins prolong gastrointestinal transit time and have an antidiarrheal effect.

Casomorphin receptor binding has been demonstrated in opiate receptor assays and bioassays. Duodenal aspirates from human volunteers given cow's milk have demonstrated the presence of several casomorphins, particularly β-casomorphin-7. Few studies have assessed the presence or action of casomorphins in humans. The ability of casein-derived opioid peptides to pass into the bloodstream is not well characterized, and is the subject of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Male or female
* Either self-described as having a strong liking for cheese, or have been following a vegan diet for a least the previous six months.

Exclusion Criteria:

* Unstable medical status
* Physical condition affecting eating behavior, digestion, or intestinal absorption
* Dairy allergy or lactose intolerance
* Pregnancy
* History of severe mental illness
* Smoking during the past six months
* Alcohol consumption of more than two drinks per day
* History of substance abuse or dependency followed by any current use
* Inordinate fear of blood draws

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
casomorphin quantification | Measurements will be collected on designated studys within 12-hour time frame

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine; Hope R Ferdowsian, MD, MPH, Study Director — Washington Center for Clinical Research
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Shah NP. Effects of milk-derived bioactives: an overview. Br J Nutr. 2000 Nov;84 Suppl 1:S3-10. doi: 10.1017/s000711450000218x. PMID 11242440
- [Background] Meisel H, FitzGerald RJ. Opioid peptides encrypted in intact milk protein sequences. Br J Nutr. 2000 Nov;84 Suppl 1:S27-31. doi: 10.1017/s000711450000221x. PMID 11242443
- [Background] Brantl V, Teschemacher H, Blasig J, Henschen A, Lottspeich F. Opioid activities of beta-casomorphins. Life Sci. 1981 Apr 27;28(17):1903-9. doi: 10.1016/0024-3205(81)90297-6. No abstract available. PMID 6265721
- [Background] Svedberg J, de Haas J, Leimenstoll G, Paul F, Teschemacher H. Demonstration of beta-casomorphin immunoreactive materials in in vitro digests of bovine milk and in small intestine contents after bovine milk ingestion in adult humans. Peptides. 1985 Sep-Oct;6(5):825-30. doi: 10.1016/0196-9781(85)90308-0. PMID 4080604
- [Background] Drewnowski A, Krahn DD, Demitrack MA, Nairn K, Gosnell BA. Taste responses and preferences for sweet high-fat foods: evidence for opioid involvement. Physiol Behav. 1992 Feb;51(2):371-9. doi: 10.1016/0031-9384(92)90155-u. PMID 1313591
- See also: Related Info — http://www.pcrm.org